CLINICAL TRIAL: NCT05284864
Title: Timing Evaluation of Stoma Closure (TIMES). Early vs Late Closure of Stoma After Rectal Cancer Surgery.
Acronym: TIMES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Blas Flor Lorente, General Surgery and Digestive System Service. Coloproctology Unit. Hospital Universitario y Politécnico La Fe. Principal Investigator, Associate Professor of Surgery. University of Valencia., Hospital Universitario La Fe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIMES
Record Dates: First submitted 2020-08-06; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Rectal Cancer; Total Mesorectal Excision; Ileostomy - Stoma; Ileostomy; Complications; Ileostomy Closure
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early stoma closure (Experimental): Stoma closure 2-3 weeks after rectal surgery.
  Interventions: Procedure: Stoma closure
- Late stoma closure (Active Comparator): Stoma closure 16-24 weeks after rectal surgery.
  Interventions: Procedure: Stoma closure

INTERVENTIONS:
Procedure: Stoma closure — Stoma closure after rectal surgery

SUMMARY:
The purpose of this study is to asses the safety and efficacy of early stoma closure (2-3 weeks after total mesorectal excision) vs late closure (16-24 weeks after mesorectal excision).

DETAILED DESCRIPTION:
Total mesorectal excision (TME) is considered the gold standard in obtaining a negative circumferential resection margin for cancers of the middle and lower third of the rectum. Despite all the oncological benefits,TME in ultra-low anterior resection carries some important drawbacks, such as a longer operative time, and its association with a higher rate of anastomotic leakage which increases in the most distal anastomoses.

Among the measures adopted to reduce mortality, the creation of protective ostomies has proven to be effective, however the protective ileostomy and its closure are not free of complications, such as dehydration and chronic kidney failure. In the investigator's country, various studies have analyzed this time to closure, being 10.8 months on average and with an increase in morbidity when closure is delayed the longest.

There are few prospective studies on the timing of stoma closure, which mainly focused on morbidity and mortality related to early closure. These studies did not demonstrate any significant negative effects on morbidity or mortality. The reason for early closure of the stoma is to reduce complications related to it. Although its true incidence is unknown, most patients have some type of stoma-related complication, which can be avoided or decreased in the case of early closure. In addition to the complications on the patient and their quality of life, the hospital costs secondary to them are not negligible.

The TIMES study ("TIMing Evaluation of Stoma closure") arises from the need to know the ideal moment for the closure of derivative stomata after rectal surgery.

Therefore, the hypothesis is that patients who undergo early ileostomy closure (at 2-3 weeks) after ultra-low anterior resection have fewer complications than patients with late ileostomy closure (4-6 months).

The main objective of this study is to analyze the morbidity and mortality associated with both early (early group, CASES group) and late closure (late group, CONTROL group) of the derivative ileosomy.

In this study, patients scheduled for temporary stoma closure after scheduled colorectal surgery will be randomized into two groups: early closure (14-21 days after surgery) or late closure (4th-6th month after surgery).

Patients will be followed from the time of study entry until 12 months after stoma closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal cancer (with / without metastasis) (with / without chemoterapy or radiotherapy)
* Patients undergoing low or ultra low anterior resection with anastomosis and stoma of protection.
* Patients with no intraoperative or postoperative complications.
* Radiological confirmation of the absence of anastomotic compilations (opaque enema or abdominal-pelvic CT scan with rectal contrast)
* Confirmation by rectoscopy of the absence of anastomotic compilations

Exclusion Criteria:

* Rectal cancer surgeries without anastomosis.
* Rectal cancer surgeries without stoma of protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine and compare morbidity and mortality rates in patients with early and late stoma closure | From rectal surgery to stoma closure surgery

SECONDARY OUTCOMES:
Determine and analyze quality of life assisted by the SF36 scale in early vs late ileostomy closure | 1 month, 6 month and 1 year after stoma closure surgery
  The SF36 is a short questionnaire with 36 items which measure eight multi-item variables: physical functioning (10 items), social functioning (two items), role limitations due to physical problems (four items), role limitations due to emotional problems (three items), mental health (five items), energy and vitality (four items), pain (two items), and general perception of health (five items). There is a further unscaled single item on changes in respondents' health over the past year. For each variable item scores are coded, summed, and transformed on to a scale from 0 (worst possible health state measured by the questionnaire) to 100 (best possible health state).

OTHER OUTCOMES:
Determine the patient's percentage with anterior resection syndrome, after early and late ileostomy closure assisted by the LARS scale. | 1 month, 6 month and 1 year after stoma closure surgery
  The LARS score has been validated and translated into several languages. By applying binomial regression on patient responses, the five issues that most bothered the patients were selected: incontinence for flatus, incontinence for liquid stool, frequency, clustering and urgency. Rating scale ranges from 0 to 42 points, and patients are classified into three groups: "no LARS" (0-20 points), "minor LARS" (21-29 points) and "major LARS" (30-42 points). According to the authors, the LARS score facilitates a fast identification of patients categorized as major LARS who will require treatment

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Complejo Hospitalario Universitario de Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital General de Elche, Elche
  - Hospital Josep Trueta, Girona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Univesitario de Salamanca, Salamanca
  - Hospital Universitari La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No